CLINICAL TRIAL: NCT00556218
Title: Feasibility Study of Meditation, Cognitive Function, and Quality of Life in Women With Breast Cancer
Brief Title: Meditation and Cognitive Function in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-0311
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Tibetan Meditation; Quality of Life; Cognitive Function; QOL
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tibetan Meditation (Other)
  Interventions: Behavioral: Tibetan Meditation Program
- No Meditation (Other)
  Interventions: Behavioral: No Meditation

INTERVENTIONS:
Behavioral: Tibetan Meditation Program — 12 sessions of Tibetan meditation (2 times a week), over a 6-week period. Each class will last about 60 minutes.
  Arms: Tibetan Meditation
Behavioral: No Meditation — No meditation; usual care.
  Arms: No Meditation

SUMMARY:
The goal of this behavioral research study is to learn if participating in a Tibetan meditation program helps to improve quality of life for women after chemotherapy and during recovery from breast cancer. Whether the meditation program helps to improve brain function and sleep quality will also be studied.

DETAILED DESCRIPTION:
Screening Tests:

During the "screening" visit, you will be asked 4 questions about your memory and concentration abilities. Based on how you score on this screening questionnaire, you may not be eligible to participate in the study even if you have already signed the informed consent form.

If you are found to be eligible for the study based on the screening questionnaire, you will complete some tests during the screening visit to check your memory and concentration. For example, you will be asked to remember a list of words and then be asked to recall them later. You will also complete questionnaires asking about your mood, quality of life, and other things like sleep, nervousness, and your experience with cancer. All together, the tests and questionnaires should take about 90 minutes to complete.

Study Groups:

You will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. People in Group 1 will take part in a Tibetan meditation program. People in Group 2 will be placed on a waiting list. They may participate in the meditation program 3 months after being enrolled in the study (when Group 1 has finished the follow-up visit).

Meditation Sessions:

If you are Group 1, you have 12 sessions of Tibetan meditation (2 times a week), over a 6-week period. You will be asked to complete a form asking about your satisfaction with the program at the start of each week. The form will take 1-2 minutes to complete.

The meditation sessions will take place at M. D. Anderson. During the meditation sessions, you will do deep breathing and visualization exercises and produce some sounds like "Ah." Each session will last about 60 minutes. One (1) or more of these meditation sessions may be videotaped by the study staff for check the quality of the sessions. Only the study staff will be able to view this videotape. All videos will be destroyed after the data is collected.

Participants in both groups will be mailed a questionnaire packet to fill out and send back (return postage will be included in the packets) at 1 month and then at the end of the meditation sessions (2 months). The questionnaires will ask about your mood, quality of life, and other things like sleeping habits and nervousness. The packet will take about 45 minutes to fill out. If you are in Group 2, you will receive packets at about the same time.

Your responses on these questionnaires will not be shared with your doctor. If you feel you need a doctor's opinion about anything that is asked in these questionnaires (for example, if you feel depressed or distressed), please contact your doctor.

Follow-up Visit:

One (1) month after the last meditation session (or at a similar time, for participants in Group 2), you will be asked to return to the clinic. You will take some tests to check your memory and concentration, similar to the tests you took at your screening visit. You will complete questionnaires asking about your mood, quality of life, and other things like sleep, nervousness, and your experience with cancer. All together, the questionnaires and tests should take about 90 minutes to complete.

Once the follow-up visit is complete, the study is over. After Group 1 has completed the follow-up visit, Group 2 will be given the option to take the meditation classes.

This is an investigational study. Up to 60 participants will be enrolled in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women with stage I - III breast cancer who have undergone chemotherapy (either neoadjuvant or adjuvant) 6 - 60 months prior to recruitment.
2. Women who report cognitive impairment since starting chemotherapy as assessed by four questions from the FACT-Cog.
3. Women must be 18 years or older.
4. Women must be able to read, write and speak English.
5. Women must be currently undergoing hormone therapy (e.g., Tamoxifen or AIs)
6. Willing to come to MDACC for the meditation sessions and assessment sessions.
7. Women must be within 2 hours driving distance of MDACC.

Exclusion Criteria:

1. Women who have a documented diagnosis of a formal thought disorder (e.g., schizophrenia) will be excluded from the study.
2. Women with metastatic disease to the brain or any past neurologic injury.
3. Women with a Mini-Mental State Examination score of 23 or below.
4. Women with recurrent cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-10-24 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Number of Eligible Women Approached Who Consented to be in Trial (Feasibility) | 2 Years
Women's Reported Satisfaction with Tibetan Meditation intervention | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org